CLINICAL TRIAL: NCT02049684
Title: SPARC: Shoulder PAtch for Rotator Cuff Tears
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: OR11/10063; 13/YH/0030 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-01-23; First posted 2014-01-30 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Massive Rotator Cuff Tears
MeSH Terms: interventions — Transdermal Patch

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Surgery
  Interventions: Procedure: Patch
- Physiotherapy

INTERVENTIONS:
Procedure: Patch
  Groups: Surgery

SUMMARY:
Rotator cuff tears (injury to the muscle or tendons which stabilise the shoulder) are one of the most common conditions affecting the shoulder. Small and medium sized rotator cuff tears can be managed with arthroscopic or keyhole surgery. Very large or massive tears are difficult to operate on and often have poor rates of healing. As a result surgeons have investigated the use of products to improve the outcome of surgery on massive tears.

The product that the investigators are currently using to try to improve the outcome of surgery for massive rotator cuff tears is called a patch. The patch provides a scaffold to support the muscles of the rotator cuff. Studies of rotator cuff surgery using similar patches have found that recovery is improved and there is a lower rate of postsurgical problems. The aim of this study is to look at whether using the patch improves pain and the clinical function of the shoulder after surgery. In addition, the investigators would like to understand how the patch works. To do this the investigators will scan (take images of) the shoulder using magnetic resonance imaging to look at the muscle damage in the shoulder before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound confirming massive rotator full thickness tear, unacceptable pain and disability following conservative treatment, or previous surgery that has failed, deltoid muscle that is functional, and compliance with post operative rehabilitation.

Exclusion Criteria:

* History of infection
* Neurological condition that affects the shoulder girdle
* Presence of rotator cuff arthropathy with stiffness
* Subjects with inability to give informed consent
* Pregnancy or lactation
* Malignancy
* Age less than 18 years
* Subjects currently participating in other research studies
* Subjects with the following contraindications to MRI scanning will not have an MR scan but may be asked to have alternative imaging, for example ultrasound:

  * Pacemakers
  * Surgical clips within the head
  * Certain inner ear implants
  * Neuroelectrical stimulators
  * Metal fragments within the eye or head
  * Pregnant or breastfeeding women

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Massive rotator cuff tear patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Change in supraspinatus, infraspinatous and subscapularis water:fat ratio | Baseline and 6 months post surgery
  Change in supraspinatus, infraspinatous and subscapularis water:fat ratio, assessed by MRI, 6 months postsurgery/ physiotherapy compared to baseline (presurgery/physiotherapy)

SECONDARY OUTCOMES:
Change in function, pain and patient satisfaction (Oxford Shoulder Score, EQ5D, Constant Score) | Baseline and 6 months post surgery
  Change in function, pain and patient satisfaction (Oxford Shoulder Score, EQ5D, Constant Score)
Change in muscle volume (MRI assessment) for the supraspinatus, infraspinatous and subscapularis | Baseline and 6 months post-surgery
  Change in muscle volume (MRI assessment) for the supraspinatus, infraspinatous and subscapularis
Change in Goutallier score of muscle atrophy and fatty infiltration (MRI assessment) for the supraspinatus, infraspinatous and subscapularis | Baseline and 6 months post-surgery
  Change in Goutallier score of muscle atrophy and fatty infiltration (MRI assessment) for the supraspinatus, infraspinatous and subscapularis

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom